CLINICAL TRIAL: NCT06056258
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Study to Evaluate the Efficacy of VL-NL-02 on Sleep and Mood.
Brief Title: A Study to Evaluate the Efficacy of VL-NL-02 on Sleep Quality.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vedic Lifesciences Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: NS/230402/ZYL/SQ
Record Dates: First submitted 2023-09-20; First posted 2023-09-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2024-01

CONDITIONS: Mood and Sleep Quality
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: randomized, double-blind, placebo-controlled trial.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VL-NL-02 (Active Comparator): Two capsules to be taken 45±10 mins before sleep (after dinner) for 21 days.
  Interventions: Dietary Supplement: VL-NL-02
- Placebo (Placebo Comparator): Two capsules to be taken 45±10 mins before sleep (after dinner) for 21 days.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: VL-NL-02 — Two capsules to be taken 45±10 mins before sleep (after dinner) for 21 days
  Arms: VL-NL-02
Dietary Supplement: Placebo — Two capsules to be taken 45±10 mins before sleep (after dinner) for 21 days
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to study the impact of VL-NL-02 in improving sleep quality, restorative sleep complaints, quality of life, stress levels, and sleep stages.

48 participants are expected to be randomized in a ratio of 1:1 to receive either VL-NL-02 or placebo and will be assigned a unique randomization code. Each group will have at least 20 completed participants after accounting for a dropout/withdrawal rate of 17%. The intervention duration for all the study participants is 21 days.

Participants will be asked to fill multiple questionnaires to assess sleep quality and mood imbalance.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged between ≥ 18 and ≤ 50 years with a moderately active lifestyle as assessed International Physical Activity Questionnaire - Short form (IPAQ - SF)
* Individuals with mild to moderate sleeping issues as assessed by an ISI score of ≥ 8 and ≤ 21
* Individuals with a history of at least 3 episodes of sleep disturbances in the last month.
* Individuals with a Fasting Blood glucose (FBG) ≤ 125 mg/dl
* All individuals who are free from use of sleeping pills for at least 4 weeks before screening
* Individuals with normal levels of laboratory parameters: Liver profile, Lipid profile and kidney profile. [Refer to section 3.7.3 for details on parameters included and reference ranges.]
* Individuals with no more than once per week use of pain-relieving medications.
* Individuals with body mass index between ≥18 and ≤ 30 kg/m2.
* Typical bedtime between 9 PM and 11 PM.
* Individuals willing to abstain from digital activity 3 hours prior to the PSG analysis
* Willing to maintain current dietary pattern, activity level, and stable body weight for the duration of the study, and refrain from any drastic lifestyle changes.

Exclusion Criteria:

* FBG > 125 mg/dl
* Individuals diagnosed with hypertension.
* Individuals having a systolic blood pressure ≥140 mm Hg and diastolic blood pressure ≥ 90 mm Hg.
* Individuals diagnosed with Type I and Type II Diabetes Mellitus.
* Sleep disorder is secondary to another health problem such as restless leg syndrome, post-operative state etc.
* Individuals diagnosed with insomnia.
* Consumption of hypnotic drugs (<3 months before inclusion)
* Individuals taking any other sleep promoting supplements and are unwilling to stop taking those supplements for the duration of the study period
* Individuals with history of sleepwalk
* Individuals who have bad dreams 2 or more times a week.
* Individuals who are inclined to the lifestyle factors - such as jet lag, night workers and rotational shift work.
* Individuals who currently, or in the past 6 months suffered from any mental-health disorder
* Individuals who were taking psychotropic medication, herbal preparation, antidepressants, steroids, antihistamines, narcotics or any other illicit drugs in the last three months.
* Individuals diagnosed with chronic medical conditions - such as heart problems, Gastro-intestinal, hepatic, respiratory, psychiatric, kidney, or cardiovascular disorder (<3 months before inclusion), and chronic pain since last 6 months.
* Recent (within 3 months before inclusion) change in lifestyle (food, sport and drug).
* Individuals who are regular smokers and/or consume any form of tobacco.
* Addiction, history of addiction, and/or substance abuse (tobacco, nicotine etc.).
* Heavy drinkers as defined by:

  1. For men, consuming more than 4 drinks on any day or more than 14 drinks/week
  2. For women, consuming more than 3 drinks on any day or more than 7 drinks/week
* Exaggerated consumption of tea (≥500 mL per day), coffee (≥400 mL per day), or energy drink (≥250 mL per day),
* Individuals on dietary supplements
* Pregnant or lactating woman,
* Lifestyle habits which would modify the wake-sleep rhythm or which was expected to be modified during the study period (e.g., night work)
* Known allergy to mushroom.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2023-12-04 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
To assess the efficacy of Vl-NL-02 on sleep quality using the Insomnia Severity Index (ISI). | Day 1 of intervention
  The Insomnia Severity Index has seven questions that indicates insomnia without clinical significance. The scores of 0-7 determines no clinically significant insomnia, 8-14 determines sub threshold insomnia, 15-21 has moderate severity which determines clinical insomnia and lastly 22-28 has severe insomnia. For each question, participant will be asked to circle or mark the number that best correlates with their sleep quality in the past two weeks. An increase in score will determine the severity of the insomnia.
To assess the efficacy of Vl-NL-02 on sleep quality using the Insomnia Severity Index (ISI). | Day 11 of intervention
  The Insomnia Severity Index has seven questions that indicates insomnia without clinical significance. The scores of 0-7 determines no clinically significant insomnia, 8-14 determines sub threshold insomnia, 15-21 has moderate severity which determines clinical insomnia and lastly 22-28 has severe insomnia. For each question, participant will be asked to circle or mark the number that best correlates with their sleep quality in the past two weeks. An increase in score will determine the severity of the insomnia.
To assess the efficacy of Vl-NL-02 on sleep quality using the Insomnia Severity Index (ISI). | Day 22 of intervention
  The Insomnia Severity Index has seven questions that indicates insomnia without clinical significance. The scores of 0-7 determines no clinically significant insomnia, 8-14 determines sub threshold insomnia, 15-21 has moderate severity which determines clinical insomnia and lastly 22-28 has severe insomnia. For each question, participant will be asked to circle or mark the number that best correlates with their sleep quality in the past two weeks. An increase in score will determine the severity of the insomnia.

SECONDARY OUTCOMES:
To assess impact of VL-NL-02 on Mood using Brief Mood Introspection Scale (BMIS) | Day 1, 11 and 22 of intervention
  It is a mood scale consisting of 16 mood adjectives to which a person responds. Four sub scores can be computed from the BMIS: Pleasant-Unpleasant, Arousal-Calm, Positive-Tired and Negative-Relaxed Mood.
To assess impact of VL-NL-02 on Dream as assessed by Dream and Sleep Emotions and Anxiety (DSEA) Questionnaire | Day 1, 11 and 22 of intervention
  The DSEA questionnaire has two subscales: Sleep anxiety and Dream emotional scale.
To assess impact of VL-NL-02 on Restorative sleep by using Restorative Sleep Questionnaire - Weekly Version (RSQ-W) questionnaire | Day 1, 11 and 22 of intervention
  RSQ-W is a validated scale for measuring refreshing quality of sleep. It has 9 items with answers scaled from 1 to 5. The questionnaire asks about how one felt after waking up and starting the day during the past seven days.
To assess impact of VL-NL-02 on Quality of life using RAND Short form (SF)-36 | Day 1, 11 and 22 of intervention
  The SF-36 includes multi-item scales to measure the following 8 dimensions (refer 15.2 for questionnaire):
  PF- Physical functioning (10 items in question 3) RP- Role limitations due to physical health problems (4 items in question 4) BP- Overall body pain (questions 7 and 8) SF- Social functioning (questions 6 and 10) MH - General mental health, covering psychological distress and well-being (5 items: questions 9 b, c, d, f and h) RE- Role limitations due to emotional problems (questions 5 a, b and c) VT- Vitality, energy or fatigue (4 items: questions 9 a, e, g and i) GH- General health perceptions (5 items: questions 1 and 11 a to d)
To assess impact of VL-NL-02 on Improvement in deep sleep and Rapid eye movement (REM) sleep stages by Polysomnography | Day 0, 10 and 21 of intervention
  Polysomnography refers to a systematic process used to collect physiologic parameters during sleep. Sleep stage scoring and detection of arousals for each 30-s epoch will be performed visually according to standard AASM procedures.
To assess impact of VL-NL-02 on Levels of salivary cortisol immediately after awakening | Day 1 and 22 of Intervention
  Normal ranges for cortisol are:
  Morning hours 8 10 a.m.: < 19.1 nmol/L (< 0.690 μg/dL) Afternoon hours 2:30-3:30 p.m.: < 11.9 nmol/L (< 0.430 μg/dL)
To assess impact of VL-NL-02 on Levels of serum serotonin | Day 1 and 22 of Intervention
  The normal range is 50 to 200 ng/mL (0.28 to 1.14 µmol/L) in healthy individuals
To assess impact of VL-NL-02 on Levels of urinary melatonin | Day 1 and 22 of Intervention
  The highest levels of melatonin are recorded from 3am onwards with a value of 47.35 pg/ml
To assess impact of VL-NL-02 on Levels of serum Brain Derived Neurotrophic Factor (BDNF) | Day 1 and 22 of Intervention

CONTACTS AND LOCATIONS:
Locations (5):
- India (5):
  - BAJ RR Hospital, Dombivali, Maharashtra
  - Surya Multispeciality Hospital, Nashik, Maharashtra
  - Sparsh Hospital, Navi Mumbai, Maharashtra
  - Dhanwantari Hospital, Pune, Maharashtra
  - Arora Allergy Asthma and Chest Care Hospital, Ajmer, Rajasthan

IPD SHARING:
Plan to Share IPD: Undecided